CLINICAL TRIAL: NCT07215416
Title: A Phase 1/2 Study of Antisense Oligonucleotide Therapy for Treatment of Ataxia-Telangiectasia
Brief Title: Safety and Efficacy of Mutation-targeted Precision Genetic Therapy for Ataxia-Telangiectasia (A-T)
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Timothy Yu (Other)
Responsible Party: Sponsor-Investigator, Timothy Yu, Physician, Department of Genetics and Genomics, Boston Children's Hospital, Associate Professor, Harvard Medical School Associate Member, Broad Institute, Boston Children's Hospital
Organization: Boston Children's Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB P00050954
Record Dates: First submitted 2025-09-10; First posted 2025-10-10 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Ataxia Telangiectasia
Keywords: Ataxia Telangiectasia; A-T; ASO; Intrathecal administration; ATM; ATIPEKSEN
MeSH Terms: conditions — Ataxia Telangiectasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Phase 1/2 Study of Antisense Oligonucleotide Therapy for Treatment of Ataxia - Telangiectasia (Experimental): Individuals with genetically confirmed, classic ataxia telangiectasia with at least one copy of the ASO-amenable ATM variant NM_000051.3:c.7865C>T;p.Ala2622Val, will receive the ASO at the same dose.
  Interventions: Drug: Antisense oligonucleotide targeting the ATM gene

INTERVENTIONS:
Drug: Antisense oligonucleotide targeting the ATM gene — Atipeksen is a fully modified PS-2'MOE splice-switching antisense oligonucleotide that is designed to restore normal splicing patterns in patients with the ATM c.7865C>T mutation.

SUMMARY:
This project aims to evaluate the safety and efficacy of precision genetic therapy for patients with Ataxia-telangiectasia (A-T), a rare neurodegenerative disease caused by mutations in the ATM gene. The investigators will conduct a clinical trial to study the safety and efficacy of intrathecal administration of atipeksen, a targeted genetic therapy that restores ATM gene function in A-T individuals bearing the recurrent ATM c.7865C>T variant. The aim of this study is to delay or forestall progression of neurologic symptoms in A-T and improving quality of life. Success will provide an empirical foundation for advancing additional precision genetic therapies for A-T and other neurodegenerative conditions.

DETAILED DESCRIPTION:
The goal of this protocol is to study the safety and efficacy of the investigational drug atipeksen, a mutation-specific antisense oligonucleotide (ASO), in individuals with ataxia telangiectasia (A-T). The first objective is to evaluate the safety of therapy with atipeksen, a 22-nucleotide oligonucleotide designed to ameliorate the effects of mis-splicing caused by a mutation in the ATM gene(NM_000051.3), c.7865C>T (p.Ala2622Val), when administered via intrathecal injection. The second objective is to determine if administration of intrathecal atipeksen can reduce or stabilize neurological decline using clinical and physiological biomarkers. The primary endpoint will be serial clinical neurologic assessments using the Ataxia-Telangiectasia Neurological Examination Toolkit (A-T NEST) and a structured version of the Ataxia-Telangiectasia Clinical Global Impression of Change (A-T CGI). Secondary endpoints will include videotaped clinical neurological examinations, movement pattern analyses using wearable actigraphy, and standard scales administered by PT, OT, and neuropsychology. Exploratory endpoints include serial brain imaging with volumetric analyses, neurofilament light chain, alpha-fetoprotein, and growth parameters.

ELIGIBILITY:
INCLUSION/EXCLUSION CRITERIA:

Who can take part:

* People with classic A-T confirmed by genetic testing
* Must have a specific ATM gene change (c.7865C>T)
* Must also have another ATM change that causes A-T

Who cannot take part:

People with health problems that make lumbar puncture unsafe:

* Blood clotting or bleeding problems
* Brain conditions raising pressure inside the head
* Serious heart or breathing problems
* Infection near the lower back

Other things doctors will check:

* Overall health and stability
* Any medicines that might cause problems
* Past difficulties with lumbar punctures
* Any other safety concerns

Ages: 0 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2035-12 (Estimated)

PRIMARY OUTCOMES:
Neurological function as measured by the AT-NEST scale | At Baseline and every 12 weeks up to ten years
  The Ataxia-Telangiectasia Neurological Examination Toolkit (AT-NEST) is a test designed specifically for people with Ataxia-Telangiectasia (A-T). It helps doctors and researchers understand how the brain and nerves are working. The test looks at six main areas:
  * Communication
  * Eye movements Ataxia (problems with balance and coordination)
  * Movement disorders
  * Muscle strength (Power)
  * Nerve function (Neuropathy) These six areas make up the "pure neuro" score, which ranges from 0 (lowest) to 100 (highest). The test also includes growth and nutrition. When these are added to the six main areas, a total "neuro-related" score is calculated, with a maximum of 114. Higher scores mean better overall performance.This test is not painful and is carried out by trained specialists who will guide you through each step.
Ataxia-Telangiectasia Structured Clinical Global Impression of Change (A-T CGI) | At Baseline and every 12 weeks up to ten years
  The Ataxia-Telangiectasia Clinical Global Impression of Change (AT-CGI) is a tool used to track how A-T progresses over time. It looks at five main areas of the disease:
  Ataxia (balance and coordination problems) Dysarthria (difficulty speaking) Repetitive movements / Dysmetria (trouble controlling movements) Movement disorders Eye movements
  Each area is scored from 0 to 4, for a total of 20 points. Higher scores mean more severe symptoms, while lower scores indicate better function.

SECONDARY OUTCOMES:
Motor performance as measured by the Bruininks-Oseretsky Test of Motor Proficiency 2nd edition | Baseline and every 6 months up to 10 years
  The Bruininks-Oseretsky Test of Motor Proficiency 2nd edition (BOT-2) is a simple way for therapists to check how your child is developing movement skills. It looks at:
  * Small hand and finger movements (fine motor)
  * How quickly and accurately hands are used (dexterity)
  * Big movements like running or jumping (gross motor)
  * How well the body works together (coordination) During the test, the child does different activities, and each one is scored. These scores are added up to give both an overall score (out of 200 points) and separate scores for each skill area. The results are then compared to what is typical for children of the same age.
Performance and goal satisfaction as measured by the Canadian Occupational Performance Measure (COPM) | Baseline and every 6 months up to 10 years
  The Canadian Occupational Performance Measure (COPM) is a test done by an occupational therapist to understand what daily activities are most important to a person and how well they feel they can do them. During the test, the person picks up to five activities they find difficult or want to improve. For each activity, they rate:
  * How well they can do it
  * How satisfied they are with their performance Both scores range from 1 to 10 (higher numbers mean better performance or more satisfaction). The scores are then averaged to see overall progress. The main goal is to track improvements over time, especially before and after a therapy or intervention.
Performance in activities of daily living as measured by the Pediatric Evaluation of Disability Inventory Computer Adaptive Test | Baseline and every 6 months up to 10 years
  The Pediatric Evaluation of Disability Inventory - Computer Adaptive Test (PEDI-CAT) is a questionnaire filled out by parents or caregivers. It helps us understand how a child is doing in everyday life. It looks at four areas:
  * Daily activities (like eating, dressing, and personal care)
  * Mobility (how a child moves around)
  * Social/cognitive (how a child plays, communicates, and learns)
  * Responsibility (how much a child can manage tasks at home or in the community) The test is "adaptive," meaning the questions change depending on how you answer, so it fits your child's abilities. Each area gets a score from 0 to 100, with higher scores meaning better functional ability.
Visual-motor function as measured by the Beery-Buktenica Developmental Test of Visual Motor Integration | Baseline and every 6 months up to 10 years
  The Beery-Buktenica Developmental Test of Visual-Motor Integration (Beery-VMI) is a test often given by occupational therapists to see how well a child's eyes and hands work together. During the test, the child copies shapes and designs that get harder as the test goes on. Sometimes the child may also be asked to find differences between pictures or match patterns. The results show:
  * A standard score with a range of 45 to 155; higher scores indicate a better performance
  * A percentile score, which shows what percentage of children the same age scored lower.
  This helps parents and therapists see how the child's coordination and fine motor skills are compared to others their age.
Neurodevelopmental function, as measured by the Leiter International Performance, third edition | Baseline and yearly up to 10 years
  The Leiter International Performance Scale-3 (Leiter-3) is a test that measures thinking and problem-solving skills. It is especially helpful for children or adults who have speech, language, or learning difficulties, or for those who do not speak English. The test looks at areas such as:
  * Problem-solving and reasoning
  * Attention and memory Visual and spatial skills (understanding shapes, patterns, and space) The results include an IQ score (higher scores mean stronger skills). Subtest scores range from 0 to 20 and composite scores range from 30 to 170; higher scores indicate a better outcome.
  This helps show how a person's thinking skills compare to others their age.
Neurodevelopmental function, as measured Wechsler Intelligence Scale for Children, fifth edition | Baseline and yearly up to 10 years
  he Wechsler Intelligence Scale for Children - Fifth Edition (WISC-V) is a test that measures different areas of a child's thinking and learning. It looks at skills such as:
  * Understanding and using language (verbal comprehension)
  * Solving puzzles and understanding visual information (visual-spatial)
  * Problem-solving and reasoning (fluid reasoning)
  * Remembering information (working memory)
  * How quickly the brain processes information (processing speed) Subtests have scaled scores with a range of 1 to 19 and composites have standard scores with a range from 45 to 155; higher scores indicate a better outcome.
  The test gives a Full Scale IQ (FSIQ) score, which shows a child's overall level of thinking skills. Higher scores mean stronger abilities.
Neurodevelopmental function, as measured by the Vineland Adaptive Behavior Scale | Baseline and yearly up to 10 years
  The Vineland Adaptive Behavior Scales, Third Edition (Vineland-3) is a test that measures how a child or adult manages everyday life skills, also called adaptive behaviors.It looks at areas such as:
  * Communication (understanding and using language)
  * Daily living skills (self-care, getting dressed, eating)
  * Socialization (interacting with others)
  * Motor skills (movement and coordination) Subtests are calculated as v-Scale scores with a possible range of 1 to 19. Composite scores are Standard Scores with a range of 20 to 140. Higher scores indicate a better outcome Growth scale values (GSVs) describe the participant's absolute level of performance on a test. Range is 10 to 220. Higher scores indicate better performance The results are turned into scores that show how well a person is functioning in daily life. Higher scores mean stronger everyday skills.
Motor performance through digital wearable actigraphs | Baseline and every 12 weeks up to 10 years
  Digital actigraphs are small motion sensors that track how a person moves during daily life. They are often used in people with movement disorders, like ataxia and ataxia-telangiectasia.
  In this study, participants will wear one sensor on the wrist and one on the ankle for one week at a time. The information collected will show how a person moves during everyday activities. These results will then be compared to others with ataxia-telangiectasia who are not receiving treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Yu, MD, PhD, Study Director — Boston Childrens Hostpital

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kim J, Woo S, de Gusmao CM, Zhao B, Chin DH, DiDonato RL, Nguyen MA, Nakayama T, Hu CA, Soucy A, Kuniholm A, Thornton JK, Riccardi O, Friedman DA, El Achkar CM, Dash Z, Cornelissen L, Donado C, Faour KNW, Bush LW, Suslovitch V, Lentucci C, Park PJ, Lee EA, Patterson A, Philippakis AA, Margus B, Berde CB, Yu TW. A framework for individualized splice-switching oligonucleotide therapy. Nature. 2023 Jul;619(7971):828-836. doi: 10.1038/s41586-023-06277-0. Epub 2023 Jul 12. PMID 37438524